CLINICAL TRIAL: NCT02482415
Title: Effects of a Psycho-educational Intervention for Family Caregivers in Palliative Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ersta Sköndal University College (Other)
Collaborators: Karolinska Institutet (Other); Linnaeus University (Other); Lund University (Other)
Responsible Party: Principal Investigator, Anette Henriksson, PhD, lecturer in Palliative Care, Ersta Sköndal University College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 130121
Record Dates: First submitted 2015-06-22; First posted 2015-06-26 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Cancer
Keywords: Palliative Care; Randomized controlled trial; Family caregivers; Intervention; Family; Intervention studies; Home Care
MeSH Terms: conditions — Neoplasms

ARMS (2):
- Intervention (Experimental): Family caregivers were invited to meet in a group for 2 hours once a week for 3 weeks. Each meeting had a specific topic presented by a health care professional of the palliative care team (physician, nurse and social worker). The meetings addressed multi-dimensional issues in dialogue with the participants. A nurse acted as group leader and participated in all meetings. The intervention included both supportive and educational components. Each meeting began with a presentation based on a specific topic (palliative care, practical care and emotional reactions). This was followed by reflection and conversation, and finally a relaxation exercise
  Interventions: Other: Psycho-educational
- Control (No Intervention)

INTERVENTIONS:
Other: Psycho-educational
  Arms: Intervention

SUMMARY:
Health care systems are increasingly using outpatient care for patients with advanced cancer disease with complex needs, limited life expectancy, and need for palliative care. Family caregivers are centrally important, but are often insufficiently prepared for the caregiving role, and experience psychological distress and physical symptoms. We hypothesize that a psycho-educational intervention during ongoing palliative care will support family caregivers' wellbeing and decrease negative consequences of caregiving.

The intervention, which has been developed in steps through a series of studies based on theoretical, methodological, and empirical work, was delivered in a group format 2013-2014. Family caregivers were invited to meet in a group for 2 hours once a week for 3 weeks. Each meeting had a specific topic presented by a member of the palliative care team (physician, nurse, and social worker). The meetings addressed multi-dimensional issues in dialogue with the participants.

The overall aim of this ongoing project is to investigate short and long-term effects of the intervention delivered by health professionals at ten specialized palliative home care units. Multiple methods are now being used, including a randomized controlled trial (RCT). In total, 270 family caregivers have been requested to answer a questionnaire at four time points: at baseline, upon completion and again 2 months after completion of the intervention, and 6 months after the patient's death. The primary outcome variable is preparedness for caregiving, and the secondary outcome variables cover aspects of wellbeing including competence and reward, caregiver burden, health, anxiety and depressive symptoms, and grief. These data will be complemented with interviews.

The project has the potential to contribute knowledge about the development of support for family caregivers, not only in specialized palliative care but also in other contexts such as elderly care and general home care services.

DETAILED DESCRIPTION:
Specific aims are to:

I) Determine the effects of the intervention upon completion, in relation to preparedness for caregiving, competence for caregiving, reward of II) Determine the effects of the intervention in a 2-month follow-up, in relation to preparedness for caregiving, competence for caregiving, reward of caregiving, health, anxiety, depressive symptoms, and caregiver burden III) Determine the effects of the intervention 6-month after the death of the patient, in relation to the family caregiver's health, anxiety, depressive symptoms and grief IV) Identify characteristics of family caregivers who do not respond to the intervention and describe support needs for these individuals V) Investigate associations between preparedness for caregiving (main outcome) and competence for caregiving, reward of caregiving, health, anxiety, depressive symptoms, caregiver burden and grief (secondary outcomes) VI) Evaluate intervention processes from the perspective of family caregivers and health care professionals VII) Investigate the influences of the caregiver intervention, for the patients with advanced cancer disease

A psycho-educational intervention was developed based on the theoretical framework of Andershed and Ternestedt relating to the principal support needs of family caregivers. The framework describes family caregivers' involvement in caregiving, and focuses on knowing, being and doing. Knowing is considered crucial for family caregivers, and is connected to an awareness of the nature of the caregiving role: knowing what to expect and what to do. Being is related to the management of one's own emotions and those of one's relative. Doing covers the practical care acts including a range of activities. It is assumed that insight will increase family caregivers' possibilities for making choices and for their involvement in caregiving.

The aim of the intervention is to increase family caregivers' feelings of preparedness for caregiving, to support their wellbeing, and to decrease negative consequences associated with caregiving. Preparedness refers to how ready family caregivers perceive they are for the tasks and demands of the caregiving role, such as providing physical care, providing emotional support and dealing with the stress of caregiving. It is suggested that preparedness could support wellbeing and protect against negative consequences in relation to caregiving. The intervention is delivered as a programme in a group format and its components, design, acceptability, feasibility and potential effects have been confirmed in a series of previous studies. During the development process, slight modifications concerning the content and structure have been done based on participant experiences.

Family caregivers were invited to meet in a group for 2 hours once a week for 3 weeks. Each meeting had a specific topic presented by a health care professional of the palliative care team (physician, nurse and social worker). The meetings addressed multi-dimensional issues in dialogue with the participants. A nurse acted as group leader and participated in all meetings. The intervention included both supportive and educational components. Each meeting began with a presentation based on a specific topic (palliative care, practical care and emotional reactions). This was followed by reflection and conversation, and finally a relaxation exercise

The intervention was conducted at ten specialized palliative home care units in the Greater Stockholm area. These settings provide palliative care mainly for patients with advanced cancer disease and complex needs and limited survival expectancy. The needs of the patients include symptom management, emotional and spiritual support, and assistance with personal nursing care.

All settings delivered 24-hours-a-day services and were staffed by multi-professional teams including physicians, nurses, social workers, occupational therapists and physiotherapists. The intervention was delivered altogether 21 times during 2013 and 2014. To ensure consistency, the content and structure of the intervention followed a manual that was developed in collaboration between researchers and staff. In order to strengthen this consistency, all team members involved in delivering the intervention participated in a 1-day workshop covering the theoretical basis of the intervention and how it should be conducted. In addition, several meetings between researchers and health care professionals were held pre-intervention, and during and after the intervention. The researchers also arranged meetings to give health care professionals from the various settings a chance to meet and share experiences related to delivering the intervention.

Both patients and family caregivers were included in the study. The inclusion criteria for patients were: being in receipt of palliative care, and having a limited life expectancy that was nevertheless assumed to be >5 weeks. Patients were not included in active data collection, but were asked to consent to the use of specific information from their medical record, including diagnosis and illness duration. Patients were also asked for approval for and preferences of which family caregiver(s) were to be asked to participate in the study. The inclusion criteria for family caregivers were: being ≥18 years old, and being able to understand and speak Swedish. All participants were consecutively approached by health care professionals and received written study information from the researchers. Family caregivers who agreed to participate were randomized to either the intervention or a control group (i.e. standard care).

In total, 270 family caregivers have been included and have been requested to answer a questionnaire to determine the effects of the intervention at four time points: at baseline, upon completion, 2 month after completion of the intervention and 6 months after the patient's death.

Inclusion and baseline assessment was completed in March 2014 with an end of intervention delivery in April 2014. The 2-month follow-up assessments for these participants were completed in June 2014. The long-term assessment may be extended since its timing is dependent on the time of death of the patient. All data collection will, however, be finalized by December 2015. Data has been collected from family caregivers, patients and health care professionals in order to evaluate the intervention and its influences as well as intervention delivery

To determine the effects of the intervention, participant assessments are made at four time points: before randomization (i.e. at baseline), upon completion of the intervention, 2 months after the intervention and 6 months after the patient's death

The questionnaire includes background characteristics such as age, sex, living conditions, level of education, relationship with the patient, marital status, financial situation, morbidity, and health care needs. It also includes scales with documented validity and reliability. The primary outcome variable is measured using the Preparedness for Caregiving Scale (PCS). The secondary outcome variables are measured using the Caregiver Competence Scale (CCS), Reward of Caregiving Scale (RCS), Caregiver Burden Scale (CBS), Health Index (HI), and Hospital Anxiety and Depression Scale (HADS). Social support is measured using the Multidimensional Scale of Perceived Social Support (MSPSS), grief is measured using the Anticipatory Grief Scale (AGS) & Texas Revised Inventory of Grief (TRIG)), and background data are assessed to identify characteristics for family caregivers who will not respond to the intervention

Interviews have been conducted with the aim to evaluate intervention processes from the perspective of family caregivers and describe influences for patients. With the aim of describing the need for support among family caregivers who do not respond to the intervention, interviews are being planned. Focus group interviews have been conducted with the aim to evaluate the intervention processes from the perspective of care professionals. The number of participants for experiential explorative studies were based on sampling principles for qualitative methods and included: 19 interviews with family caregivers 25 Health care professionals. Approximately 20 interviews with family caregivers who do not respond to the intervention will be held.

Data analysis To secure the statistical power for the regression analyses, sample size calculations were made. A sample of 110 would be sufficiently large to detect a medium effect size.

Descriptive statistics, χ2 statistics for categorical variables, and Student's t-test (unpaired) for continuous data (or equivalent non-parametric tests) were used to describe the characteristics of the participants and to compare the intervention and control group at baseline. Due to violations of the assumption of independence multiple linear regression analysis based on robust variance estimates was conducted to test the short and longer-term effects of the intervention (at baseline, upon completion of the intervention and two months following the intervention) and 6 months after the patient's death.

Participants from the intervention group will be categorized into those who demonstrate improvement and those who do not and descriptive statistics will be used to identify characteristics associated with this distinction. Age, sex, living conditions, educational level, relation to the patient, marital status, financial situation, morbidity, health care needs, social support, and anticipatory grief will be included as predictor variables.

Multiple linear regression analyses will be used to investigate the association between study outcome variables.

Analyses of interviews and focus group data were conducted with interpretive descriptive analysis during data Collection.

Ethical considerations A guiding ethical principle is not to harm the study participants, whether they participate in the intervention or in the control group. We have considered that answering the questionnaire and participating in the interviews may be associated with strong emotions. In addition, we have considered the stressful situation for caregivers. For this reason, the written and oral information emphasizes the voluntary nature of participation and the right to withdraw from the study at any time point. Ethics approval for the project and the extended project has been obtained from the regional ethical review board in Stockholm (2012/377-31, 2012/2191-32, 2013/934-32).

Significance and clinical relevance The Project is based on an RCT design contributing to high evidence value results. It was hypothesized that a psycho-educational intervention delivered by health care professionals during ongoing palliative care would support family caregivers of patients with advanced cancer disease, sustain their wellbeing and decrease the negative consequences of caregiving. The project will expand the knowledge about short and long-term effects as well as intervention processes and influences of the intervention from the perspective of family caregivers, health care professionals and patients. The studies can thereby prepare for implementing the intervention in clinical settings. The intervention was planned, designed and conducted in cooperation with the health care professionals who were responsible for its delivery at ten specialized palliative home care units. This will further facilitate implementation of the intervention and research results - not only at the study settings, but also at other specialized palliative home care units. The RCT design should enhance the generalizability of the results and make the intervention applicable to implement as a tool in clinical practice. The project also has the potential to generate results that will contribute to the development of support for family caregivers in other contexts, for example elderly care and general home care services. Overall, the project has a potential to contribute to the body of knowledge about intervention development, delivery, and evaluation during ongoing palliative care.

ELIGIBILITY:
Inclusion Criteria:

* Being family caregiver to a person in specialized palliative home care,
* Over the age of 18, and
* Able to read and understand Swedish.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in the PCS 5 weeks and 13 weeks after baseline | Baseline, 5 weeks, 13 weeks
  The PCS is designed to measure caregivers' perceived readiness to provide care in real time. It consists of eight items answered on a five-point Likert-type response scale ranging from 'not at all prepared' (0) to 'very well prepared' (4) with a total score ranging from 0-32.
TRIG | 6 months after the patient's death
  TRIG measures complicated grief on a 5 Point likert type scale ranging from 1 (Completely true) to 5 (Completely false).

REFERENCES:
- [Derived] Holm M, Arestedt K, Carlander I, Wengstrom Y, Ohlen J, Alvariza A. Characteristics of the Family Caregivers Who Did Not Benefit From a Successful Psychoeducational Group Intervention During Palliative Cancer Care: A Prospective Correlational Study. Cancer Nurs. 2017 Jan/Feb;40(1):76-83. doi: 10.1097/NCC.0000000000000351. PMID 26925988